CLINICAL TRIAL: NCT00067054
Title: VRC 200: A Multicenter Specimen Collection Protocol to Obtain Human Biological Samples for Research Studies
Brief Title: Apheresis and Specimen Collection Procedures to Obtain Plasma, Peripheral Blood Mononuclear Cells (PBMCs) and Other Specimens for Research Studies
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030263; 03-I-0263
Record Dates: First submitted 2003-08-08; First posted 2003-08-11 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Sample Collection
Keywords: Volunteer; Plasmapheresis; Leukapheresis; Immunology; Leukocyte; Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Sample collection only

SUMMARY:
This study collects specimens from volunteers for use in studies by NIAID's Vaccine Research Center. A number of different types of specimens or samples can be collected, including blood, urine, body fluids or secretions, skin swabs, or skin biopsies. The samples are used for medical research, including the study of HIV, hepatitis, and other diseases; immune system responses, such as responses to vaccinations or infections; and for research on vaccine development.

Blood samples may be collected either by ordinary blood drawing (phlebotomy) or by apheresis, a procedure for collecting a larger quantity of blood cells or plasma than would be possible through simple blood drawing. For this procedure, the participant lies on a recliner or couch. Blood is removed through a needle in the vein of one arm and spun in a machine that separates out the desired component (plasma or white blood cells). The remainder of the blood is returned either through the same needle or through a needle in the other arm. The procedure takes about 1 to 3 hours.

Volunteers who are 18 years of age and older, including participants in other NIH research protocols, may be eligible. Individuals who have a condition that the research staff considers a reason not to make a sample donation will be excluded from the study.

Participants may have only one sample collected or may be asked to undergo repetitive sample collection procedures, depending upon the requirements of the particular research project for which the samples are being collected. Each individual's enrollment is for a 1-year period, which can be extended.

DETAILED DESCRIPTION:
Study Description:

This protocol is designed to collect human specimens, such as blood, mucosal secretions, skin swabs, skin biopsy, or body fluids to support medical research. These samples will be used by researchers in their work on the development of vaccines and monoclonal antibodies, to study the correlates of immunity related to infectious diseases and allergies, and in laboratory work related to the development and/or validation of immunological and other relevant assays. Standard phlebotomy and apheresis procedures will be utilized to safely obtain necessary quantities of blood and cells.

Objectives:

To obtain human biological specimens such as blood (via phlebotomy), plasma or peripheral blood mononuclear cells (PBMC) samples (via apheresis), mucosal secretions, skin swabs, body fluids, and skin biopsy to support medical research.

Study Population:

Children, ages 3-17 years and adults, ages 18 years and older.

Protocol Plan:

Participants, including healthy volunteers and patients with an infection or with an allergic or autoimmune condition who consent to participate in this study, will undergo standard medical procedures to obtain biological specimens. Samples may be collected at clinic visits by study staff, at outside laboratories or healthcare providers, or at home by the participant and shipped to the NIH by the participant.

Study Duration:

Individual participants may donate samples as often as permitted by their institution s guidelines. The IRB-approved protocol will remain open and undergo annual continuing review by the IRB.

Endpoints:

There are no specific endpoints in this study, as samples are collected for investigations conducted in research laboratories to address questions related to immunity and vaccine and monoclonal antibody development. Therefore, there is no analysis plan for this protocol. This protocol will be conducted in accordance with Good Clinical Practices for human research solely for the purpose of obtaining samples for research laboratories. Samples will be identified only by a participant identification number. Non-personally identifying information that will be linked to a participant ID only, such as demographic information, aspects of the medical history, laboratory parameters, recent immunizations or medications, genetic tests, and other medical information, may be provided to researchers if needed to support the objectives of the laboratory research.

ELIGIBILITY:
* INCLUSION CRITERIA FOR ADULT PARTICIPANTS:

A participant must meet all the inclusion criteria, as follows:

1. Age 18 years or older
2. Able and willing to complete the informed consent process
3. Willing to provide blood or other samples that will be stored indefinitely and used for future research
4. Able to provide proof of identity to the acceptance of the clinician completing the enrollment process; when informed consent is obtained by telephone or a telehealth visit, the investigator obtaining consent will also confirm proof of identity.

INCLUSION CRITERIA FOR CHILDREN:

1. Children aged 3 to 17 years inclusive, and at least 12 kg in weight.
2. Capability of the legal adult guardian of the child to understand and comply with the planned study procedures.
3. Capability of the legal adult guardian of the child to provide written informed consent.
4. Willing to have blood drawn or collection of urine, fecal samples, oral secretions, or swabs of mucosa that will be stored indefinitely and used for future research.
5. The legal adult guardian of the children can provide proof of identity for the child and for themselves to the satisfaction of the clinician completing the enrollment process.

EXCLUSION CRITERIA FOR ALL PARTICIPANTS:

A participant will be excluded from protocol participation if there is presence of a condition that the attending physician considers to be a contraindication to the specimen collection procedures.

EXCLUSION CRITERIA FOR CHILDREN ONLY

1. Acute or chronic illness that, in the opinion of the investigator or designee, precludes participation in the study.
2. Factors related to the legal guardian that, in the judgment of the investigator or designee, may affect the objective decision-making of the legal guardian.

SKIN BIOPSY ELIGIBILITY CRITERIA FOR ADULTS ONLY:

The skin biopsy eligibility includes the following:

1. Age 18 years or older
2. No known allergies to the local anesthetic to be used
3. No history of keloid formation
4. No known coagulation disorders
5. Not pregnant or breast feeding

APHERESIS ELIGIBILITY CRITERIA FOR ADULTS ONLY:

* To undergo an apheresis procedure, a participant must have no medical contraindications. All apheresis procedures performed under this protocol are solely for research purposes.
* Participants involved in an active clinical research protocol may participate in the apheresis protocol if the total amount of blood drawn does not exceed NIH guidelines or a site's institutional guidelines. A study clinician will complete a checklist for apheresis eligibility before referring a participant for apheresis.
* At the NIH, prior to the scheduled procedure, the participant must have a venous assessment performed by apheresis staff to determine suitability for apheresis.

For Healthy Volunteers:

A healthy volunteer must meet all the following criteria prior to the procedure:

1. Age 18 years or older
2. Afebrile (temperature <= 37.50 degrees C)
3. Weight >=110 pounds
4. Adequate bilateral antecubital venous access
5. Hemoglobin >= 12.5 g/dL for women; >= 13.0 g/dL for men within 56 days prior to apheresis procedure.
6. Platelets > 150,000 K/uL within 56 days prior to apheresis procedure.
7. No cardiovascular instability as indicated by a) history of medically significant cardiac arrhythmia within the last 12 months, or b) ischemic cardiovascular disease within the last 12 months, or c) heart rate outside of the 50-100 beats/minute interval (on 3 successive readings), or d) blood pressure greater than 180 mmHg (systolic) or 100 mmHg (diastolic) on 3 successive readings
8. No current lung or kidney disease
9. No known coagulation disorder
10. No sickle cell disease
11. No active or chronic hepatitis
12. No intravenous injection drug use in the past 5 years
13. Not breast feeding
14. Negative beta-human chorionic gonadotropin (beta-HCG) pregnancy test (urine or serum) performed by a VRC study clinician within 72 hours prior to the apheresis procedure

Patients with an Infectious Disease:

A patient with an infectious disease must meet all the following criteria:

1. Age 18 years or older
2. Weight >= 110 pounds
3. Afebrile (temperature <= 37.5 degrees C)
4. Adequate bilateral antecubital venous access
5. No cardiovascular instability as indicated by a) history of medically significant cardiac arrhythmia within the last 12 months, or b) ischemic cardiovascular disease within the last 12 months, or c) heart rate outside of the 50-100 beats/minute (on 3 successive readings), or d) blood pressure greater than 180/100 mmHg (on 3 successive readings)
6. No current lung or kidney disease
7. No known coagulation disorder
8. No receipt of clotting factor concentrates in the past 5 years
9. Hemoglobin >= 9.0 g/dL within 56 days prior to apheresis procedure
10. Platelets >= 50,000 K/uL within 56 days prior to apheresis procedure
11. White Blood Cell WBC >= 2.0 K/uL within 56 days prior to apheresis procedure
12. Not breast feeding
13. Negative beta-human chorionic gonadotropin (beta-HCG) pregnancy test (urine or serum) performed by a VRC study clinician within 72 hours prior to the apheresis procedure

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants may be individuals participating solely in this protocol or may be individuals in other VRC studies from whom more cells are needed for research than can be collected by routine phlebotomy.At the VRC site, NIH employees and members of their immediate families may participate in this protocol. The UPR MSC site will only enroll participants from the community. Children are not eligible to participate in this clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2003-09-10 (Actual)

PRIMARY OUTCOMES:
Sample collection only | end of study
  This protocol does not have an analysis primary outcome measure, but rather will be conducted in accordance with Good Clinical Practices for human research solely for the purpose of obtaining samples for research laboratories. Samples will be identified only by protocol identification number. Participant data, such as demographic information, aspects of medical history, laboratory parameters, recent immunizations or medications, HLA type, genetic tests and other medical information may be provided (identified by study number, but not subject name) to researchers if needed to support the objectives of the laboratory research.

CONTACTS AND LOCATIONS:
Overall Officials: Lesia K Dropulic, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - EvergreenHealth Medical Center, Kirkland, Washington
- University of Puerto Rico Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Background] Strauss RG, Maguire LC, Koepke JA, Thompson JS. Effect of intermittent-flow centrifugation leukapheresis on donor leukocyte counts. Acta Haematol. 1980;63(3):128-31. doi: 10.1159/000207383. PMID 6769278
- [Background] Heal JM, Horan PK, Schmitt TC, Bailey G, Nusbacher J. Long-term follow-up of donors cytapheresed more than 50 times. Vox Sang. 1983;45(1):14-24. doi: 10.1111/j.1423-0410.1983.tb04118.x. PMID 6410585
- [Background] Braine HG, Elfenbein GJ, Mellits ED. Peripheral blood lymphocyte numbers, lymphocyte proliferative responses in vitro, and serum immunoglobulins in regular hemapheresis donors. J Clin Apher. 1985;2(3):213-8. doi: 10.1002/jca.2920020302. PMID 4030708
- [Derived] Zhou T, Teng IT, Olia AS, Cerutti G, Gorman J, Nazzari A, Shi W, Tsybovsky Y, Wang L, Wang S, Zhang B, Zhang Y, Katsamba PS, Petrova Y, Banach BB, Fahad AS, Liu L, Acevedo SNL, Madan B, de Souza MO, Pan X, Wang P, Wolfe JR, Yin M, Ho DD, Phung E, DiPiazza A, Chang L, Abiona O, Corbett KS, DeKosky BJ, Graham BS, Mascola JR, Misasi J, Ruckwardt T, Sullivan NJ, Shapiro L, Kwong PD. Structure-Based Design with Tag-Based Purification and In-Process Biotinylation Enable Streamlined Development of SARS-CoV-2 Spike Molecular Probes. SSRN [Preprint]. 2020 Jul 21:3639618. doi: 10.2139/ssrn.3639618. PMID 32742241
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-I-0263.html